CLINICAL TRIAL: NCT05911139
Title: Influence of General Anesthesia on the Dynamic Changes in Brain Damage Markers During and After Craniosynostosis Operations in Infancy
Acronym: TAnBrainDam
Status: Enrolling by invitation | Type: Observational
Sponsor: Comenius University (Other)
Responsible Party: Sponsor
Other Study IDs: EK2/2022/2405; 1/0564/23 (Other Grant/Funding Number: VEGA)
Record Dates: First submitted 2023-06-12; First posted 2023-06-20 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Craniosynostosis; Anesthesia
Keywords: anesthesia; children; neurotoxicity; neuron specific enolase; S100B protein; neurofilament light chain
MeSH Terms: conditions — Craniosynostoses; Neurotoxicity Syndromes; Charcot-Marie-Tooth disease, Type 1F

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Biospecimen Retention: Samples Without DNA — blood sampling - before anesthesia, at the end of anesthesia and 48 hours after the end of anesthesia - determination of S100B protein level
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- pediatric patients: Patients indicated for surgical treatment of single-layer craniosynostosis will be selected for the study, anticipated 15 patients per calendar year

SUMMARY:
The issue of anesthetics neurotoxicity is one of the most discussed topics in pediatric anesthesiology, thus it opens the question of the safety of commonly used anesthetics in the pediatric patient. Preclinical studies have shown that anesthetics can have a toxic effect on the maturing brain of pups and cause cognitive impairment. In human medicine, the influence of anesthetics is studied by monitoring the psychomotor development of children who have undergone surgery under general anesthesia. Some work deals with laboratory evidence of brain damage due to general anesthesia, but none of the work deals with the observation of markers of brain damage in infants. The aim of this work is to examine the dynamics of changes in the concentrations of selected markers of brain damage in craniosynostosis operations under general anesthesia in infants in order to optimize perioperative management and the correct timing of surgery.

DETAILED DESCRIPTION:
More than twenty years ago, experimental work found that anesthetics can be toxic to the maturing brain of animal pups and cause cognitive impairment (Ikonomidou, 1999). The presented evidence suggested that the action of commonly used anesthetics triggers biochemical and morphological changes in immature neurons, which ultimately lead to their extinction (Creeley, 2013; Liu, 2012; Brambrink, 2010). Recent clinical studies have shown that general anesthesia can also have a negative effect on a child's cognitive functions (DiMaggio, 2017; Bong, 2013; Naumann, 2012; Flick, 2011). In another published study, it was found that the effect of general anesthesia in younger children leads to a more significant increase in markers of brain damage, neuron-specific enolase (NSE) and S100B protein (S100B), compared to older children (Stojanovic Stipic, 2017). It has also been shown, that the level of neurofilament light chain (NfL), a biomarker of axonal damage found in wide variety of neurological disorders (Khalil, 2018), is increased in adult patient's blood after anesthesia (Evered, 2018). Knowing the dynamics of brain damage markers can help optimize perioperative management and consideration of postponing the consider postponing surgery until later in childhood.

The aim of the submitted project is:

1. To determine the dynamic changes in the concentration of selected markers of brain damage (NSE, S100B and NfL) during inhalation anesthesia in infants.
2. To determine the dynamic changes in the concentration of these markers depending on:

   A) age of the child B) duration of general anesthesia C) type of operation (open cranioplasty versus endoscopic cranioplasty)
3. Assessment of psychomotor development in the preoperative and postoperative period with an interval of 1 year after the operation and in the 36th month of the child's life.
4. Analysis of the relationship between changes in psychomotor development and changes in the concentration of brain damage markers.
5. Publication and implementation of the results into clinical practice.

Main benefit:

1. Optimization of surgical treatment of craniosynostosis with regard to minimizing the neurotoxic effect of anesthesia.

   Secondary benefits:
2. Determining the dynamics of changes in the values of selected markers of brain damage under general anesthesia in craniosynostosis operations. Monitoring the relationship of selected parameters (length of anesthesia, patient age, weight, sex, type of surgical correction (endoscopic vs open), type of craniosynostosis, blood loss + correction and side reactions to changes in brain damage markers (NSE, S100B and NfL)).

   Despite the fact that the investigators do not yet have clear results of the study, or a clear consensus of professional societies, the investigators assume that general anesthesia, especially repeated or long-term, can affect the maturing central nervous system of the child. The assumption is that due to the vulnerability of the brain, the increase in markers will be higher in the younger age of the child (endoscopic cranioplasty). European anesthesia societies do not share the FDA's full view. They mainly disagree with the insufficiently substantiated determination of the age limit of 3 years and the duration of general anesthesia of more than 3 hours as a risk factor increasing the incidence of neurotoxic damage. To date, no work has been published to monitor markers of brain damage in infants under general anesthesia.
3. To help in the future specify the optimal perioperative management, the method of anesthesia and the appropriate timing of the surgical procedure in order to consider postponing it to a later age of the child and at the same time to avoid unnecessary postponement of surgical procedures.

Description of the work plan:

1. Patient recruitment, preoperative preparation

   * Prospective recruitment of patients indicated for surgical treatment of single-stage craniosynostoses at National Institute of children diseases (NICHD) Bratislava. Surgical treatment will be performed according to conventional indications (endoscopic correction in patients under 6 months of age, open correction in patients older than 6 months). Estimated number of operated patients 15 during 1 year.
   * Each child will be examined by a neurologist before and after the operation, the child's psychomotor development will be examined preoperatively (Bayley scale - Bayley III)
   * Children with ASA 1 - 2 ( ASA Physical Status Classification System), without neurological deficit, without associated diseases will be included in the group. The child's parents will sign the informed consent
2. Surgical performance under general anesthesia and perioperative marker collection

   * The operation will be performed by one surgeon and three pediatric anesthesiologists. General anesthesia will be inhaled (Sevoflurane / 02 / air opioid).
   * Each patient will have recorded monitoring parameters (length of anesthesia, patient's age, weight, sex, type of surgical correction (endoscopic vs open), type of craniostenosis, perioperative blood loss + correction
   * The concentration of markers of brain damage will be recorded immediately after the start of general anesthesia, at the end of anesthesia, 48 hours after the end of anesthesia.

Postoperative follow-up

* Monitoring the relationship between changes in brain damage markers and changes in psychometrical development (PMV) (Bayley scale - Bayley III) one year after surgery and at the age of 36 months.
* Monitoring of the child at the neurosurgical outpatient clinic one month after the operation, 6 months after the operation, 1 year after the operation, at the 36th month of the child's life.

In the second and third stages /t.j. in the second and third year of the project/

1. Patient recruitment will continue.
2. Surgical treatment of craniosynostosis under general anesthesia will continue.
3. Follow-up of patients enrolled in the study will continue (monitoring the relationship between changes in brain damage markers and changes in psychometrical development (PMV) (Bayley scale) one year after surgery and at the age of 36 months).

Preoperative examinations will be coordinated by a participating neurosurgeon and anesthesiologist. Surgical intervention and perioperative examinations will be coordinated by the participating neurosurgeon.

Type of surgery. The study will use two surgical techniques: endoscopic cranioplasty and open cranioplasty.

* General anesthesia. The operation will be performed under inhalation general anesthesia (Sevoflurane / O2 / air in combination with the opioid Sufentanyl) with strict monitoring of the patient's vital signs.
* Perioperative sampling, data collection. For each patient, the patient's age, weight, sex, length of anesthesia, type of surgical correction (endoscopic vs. open), type of craniosynostosis (single suture), blood loss + correction will be recorded. Immediately after the introduction of general anesthesia, blood samples will be taken to determine NSE, S100B and NfL. Sampling will be performed regularly at hourly intervals for a control examination of acid-base balance and ionogram in order to exclude other possible factors that have a negative effect on the central nervous system.

Postoperative follow-up.

* Two postoperative blood samples will be performed to determine NSE, S100 and NfL in order to determine the further dynamics of the parameters, 1) immediately after the end of anesthesia and 2) 48 hours after anesthesia.
* On the assessment of the child's psychomotor development (PMV) (Bayley III Bayley scale) one year after surgery and at the age of 36 months.

Postoperative examinations will be coordinated by a participating neurosurgeon. Evaluation and publication of results.

* Blood biomarker levels (NSE, S100 and NfL) evaluated using standard statistical methods
* Changes in PMV using the Bayley - III method one year after surgery and at the age of 36 months.
* Based on the results, a recommendation for clinical practice will be developed.

Social and other benefits and commercial use of project outputs. The social benefits of the project result from its scientific and medical outputs. The investigators do not yet have definitive results from clinical trials or a clear consensus of professional anesthesiology societies regarding the possible neurotoxicity of anesthetics, but the investigators nevertheless assume that general anesthesia, especially long-term anesthesia, has a negative effect on a child's developing brain. A large number of procedures cannot be postponed, but it is really necessary to pay great attention to a thorough indication of the operation or examination under general anesthesia and analgesia. When indicating anesthesia, it is necessary to keep in mind the fundamental, still debated discrepancy between the degree of neurotoxicity of general anesthetics and the possible consequences of insufficient or no analgesia and anesthesia. Although recent studies suggest that a single general anesthesia (lasting less than 3 hours) is unlikely to affect a child's behavior or learning, it is really important not to underestimate the issue of neurotoxicity and to consider whether all imaging and surgical procedures under general anesthesia or analgesia it is really necessary to realize it by the age of three. Before each anesthesia, the investigators should evaluate the benefits of anesthesia against the potential risks, especially if the procedures are longer than 3 hours or repeated procedures in children under three years of age. The aim of this project is to monitor the dynamics of changes in brain damage markers in infants during surgical procedures, when general anesthesia lasts on average longer than 3 hours. This is the first project that does not only deal with the observation of psychomotor development of children under the influence of long-term general anesthesia. Several aspects of this project have not yet been published and there is a high presumption of obtaining original results.

ELIGIBILITY:
Inclusion Criteria:

* Patients indicated for surgical treatment of single-layer craniosynostosis will be selected for the study. Surgical treatment will be performed according to conventional indications (endoscopic correction in patients under 6 months of age, open correction in patients older than 6 months) under general anesthesia. ASA 1 - 2. The signing of informed consent to inclusion in the study is also a condition. In the preoperative period, the investigators will assess the achieved developmental level of the child using the Bayley scale (Bayley - III).

  * The child's parents will sign an informed consent to be included in the study.

Exclusion Criteria:

* Patients with comorbidities, syndromic craniosynostosis will be excluded from the study.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Prospective recruitment of patients indicated for surgical treatment of single-stage craniosynostoses at NUCHD Bratislava. Surgical treatment will be performed according to conventional indications (endoscopic correction in patients under 6 months of age, open correction in patients older than 6 months).
Sampling Method: Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Blood biomarker level of neuron-specific enolase (NSE) | 48 hours
  Three determinations of the level of NSE- 1, Immediately after the introduction of general anesthesia; 2, immediately after the end of anesthesia; 3, 48 hours after anesthesia
Blood biomarker level of protein S100 | 48 hours
  Three determinations of the level of protein S100- 1, Immediately after the introduction of general anesthesia; 2, immediately after the end of anesthesia; 3, 48 hours after anesthesia
Blood biomarker level of neurofilament light chain (NfL) | 48 hours
  Three determinations of the level of NfL, Immediately after the introduction of general anesthesia; 2, immediately after the end of anesthesia; 3, 48 hours after anesthesia

SECONDARY OUTCOMES:
child's psychomotor development (PMV) | 36 months
  Assessment of the child's psychomotor development (PMV) (Bayley III Bayley scale) one year after surgery and at the age of 36 months.

OTHER OUTCOMES:
other parameters- age | 1 hours
  Patient's age in months in time of surgery
other parameters- weight | 1 hour
  Patient's weight in centimeters
other parameters- sex | 1 hour
  Patient's sex (man or women)
other parameters- length of anesthesia | 4 hours
  Patient's length of anesthesia
other parameters- type of surgical correction | 1 hours
  Patient's type of surgical correction (endoscopic vs. open)
other parameters- blood loss | 1 hours
  Patient's blood loss during surgery in milliliters

CONTACTS AND LOCATIONS:
Locations (1):
- Department of paediatric anaesthesiology and intensive medicine, Bratislava, Slovakia

REFERENCES:
- [Background] McGuigan S, Evered L, Scott DA, Silbert B, Zetterberg H, Blennow K. Comparing the effect of xenon and sevoflurane anesthesia on postoperative neural injury biomarkers: a randomized controlled trial. Med Gas Res. 2022 Jan-Mar;12(1):10-17. doi: 10.4103/2045-9912.324591. PMID 34472497
- [Background] Khalil M, Teunissen CE, Otto M, Piehl F, Sormani MP, Gattringer T, Barro C, Kappos L, Comabella M, Fazekas F, Petzold A, Blennow K, Zetterberg H, Kuhle J. Neurofilaments as biomarkers in neurological disorders. Nat Rev Neurol. 2018 Oct;14(10):577-589. doi: 10.1038/s41582-018-0058-z. PMID 30171200
- [Background] Stojanovic Stipic S, Carev M, Bajic Z, Supe Domic D, Roje Z, Jukic A, Stipic T. Increase of plasma S100B and neuron-specific enolase in children following adenotonsillectomy: a prospective clinical trial. Eur Arch Otorhinolaryngol. 2017 Oct;274(10):3781-3788. doi: 10.1007/s00405-017-4698-1. Epub 2017 Aug 7. PMID 28785895
- [Background] Flick RP, Katusic SK, Colligan RC, Wilder RT, Voigt RG, Olson MD, Sprung J, Weaver AL, Schroeder DR, Warner DO. Cognitive and behavioral outcomes after early exposure to anesthesia and surgery. Pediatrics. 2011 Nov;128(5):e1053-61. doi: 10.1542/peds.2011-0351. Epub 2011 Oct 3. PMID 21969289
- [Background] Bong CL, Allen JC, Kim JT. The effects of exposure to general anesthesia in infancy on academic performance at age 12. Anesth Analg. 2013 Dec;117(6):1419-28. doi: 10.1213/ANE.0b013e318299a7c2. PMID 24132012
- [Background] Brambrink AM, Evers AS, Avidan MS, Farber NB, Smith DJ, Zhang X, Dissen GA, Creeley CE, Olney JW. Isoflurane-induced neuroapoptosis in the neonatal rhesus macaque brain. Anesthesiology. 2010 Apr;112(4):834-41. doi: 10.1097/ALN.0b013e3181d049cd. PMID 20234312
- [Background] Liu F, Patterson TA, Sadovova N, Zhang X, Liu S, Zou X, Hanig JP, Paule MG, Slikker W Jr, Wang C. Ketamine-induced neuronal damage and altered N-methyl-D-aspartate receptor function in rat primary forebrain culture. Toxicol Sci. 2013 Feb;131(2):548-57. doi: 10.1093/toxsci/kfs296. Epub 2012 Oct 11. PMID 23065140
- [Background] Ikonomidou C, Bosch F, Miksa M, Bittigau P, Vockler J, Dikranian K, Tenkova TI, Stefovska V, Turski L, Olney JW. Blockade of NMDA receptors and apoptotic neurodegeneration in the developing brain. Science. 1999 Jan 1;283(5398):70-4. doi: 10.1126/science.283.5398.70. PMID 9872743